CLINICAL TRIAL: NCT06240507
Title: Comparison of Ultrasound-guided Posterior Tibial Nerve Pulsed Radiofrequency and Fluoroscopy-guided Intralesional Radiofrequency Thermocoagulation in the Treatment of Painful Calcaneal Spur and Plantar Fasciitis
Brief Title: Posterior Tibial Nerve PRF vs Intralesional RFT for Painful Calcaneal Spur and Plantar Fasciitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Damla Yürük, Supervisor Investigator, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PTN PRF vs intralesional RFT
Record Dates: First submitted 2024-01-26; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Heel Spur; Plantar Fascitis
Keywords: Pulsed Radiofrequency Treatment; Ultrasonography; Fluoroscopy; Tibial Nerve
MeSH Terms: conditions — Heel Spur

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pulsed radiofrequency group (Active Comparator): posterior tibial nerve pulsed radiofrequency for painful calcaneal spur and plantar fasciitis
  Interventions: Procedure: ultrasound-guided posterior tibial nerve pulsed radiofrequency
- radiofrequency thermocoagulation group (Active Comparator): intralesional radiofrequency thermocoagulation for painful calcaneal spur and plantar fasciitis
  Interventions: Procedure: fluoroscopy-guided intralesional radiofrequency thermocoagulation

INTERVENTIONS:
Procedure: ultrasound-guided posterior tibial nerve pulsed radiofrequency — The posterior tibial nerve (PTN) was identified with a 5-12 MHz linear ultrasonography (US) probe at the level of the medial malleolus, where it runs posterior to the posterior tibial artery. Using the in-plane technique, a 22-gauge, 10-cm radiofrequency cannula was inserted under US guidance and advanced until the tip was adjacent to the nerve. Pulse radiofrequency was applied at 42°C for 240 s with a pulse width of 20 ms
  Arms: pulsed radiofrequency group
Procedure: fluoroscopy-guided intralesional radiofrequency thermocoagulation — The painful heel and calcaneal spur were visualized under lateral fluoroscopy. A 22-gauge, 10-cm radiofrequency cannula was inserted and advanced until the needle tip reached the calcaneal spur tip. When the needle tip contacted the spur, local anesthetic was administered through the cannula and radiofrequency ablation was performed at 80°C for 90 s.
  Arms: radiofrequency thermocoagulation group

SUMMARY:
This study aims to compare the efficacy of ultrasound (US)-guided posterior tibial nerve pulsed radiofrequency (PTN PRF) and fluoroscopy (FL)-guided intralesional radiofrequency thermocoagulation (RFT) for the treatment of painful calcaneal spur and plantar fasciitis refractory to conservative treatments. For this evaluation, a numerical rating (NRS) and the American Orthopedic Foot and Ankle Society (AOFAS) ankle hindfoot scores will be used before and after both interventions.

DETAILED DESCRIPTION:
Painful calcaneal spurs (PCS) and plantar fasciitis (PF) are common foot conditions affecting approximately 10-15% of the population. These conditions can cause severe heel pain and disability, affecting the patients' quality of life and productivity.

Treatment of these conditions is complex and sometimes resistant to conventional therapies, such as rest, ice, stretching, orthotics, and anti-inflammatory drugs. Some studies have shown that conservative treatments can improve PCS and PF symptoms within 12 months. However, if conservative treatments fail, interventional procedures such as corticosteroid injections, radiofrequency ablation, or surgery may be used on the PCS and surrounding nerves.

PRF and RFT are two modalities of thermal ablation that can be used to treat chronic pain conditions. PRF delivers short bursts of high-voltage electrical current to the target nerve, creating a non-thermal effect that modulates the transmission of pain signals. RFT delivers a continuous current that heats the target tissue, causing coagulation, and can promote thinning of hard tissues, such as calcaneal spurs and plantar fascia. The PTN is a branch of the sciatic nerve that provides sensory and motor innervation to the heel and sole of the foot, where calcaneal spurs and PF occur. The advantage of the PTN over its smaller branches is that it can be visualized and targeted using US. FL can visualize PCS.

US-guided PTN PRF and FL-guided intralesional RFT for pain management in PCS and PF have been used in a limited number of studies; however, no studies have compared their efficacy and adverse event rates.

The primary aim of this study was to compare the efficacy of these two treatment modalities. The secondary aim was to determine the incidence of adverse events associated with US-guided PTN PRF and FL-guided intralesional TRF treatment. A total of at least 46 patients, 23 patients in each group, will be enrolled for comparison. NRS, and AOFAS scores before, 1 month, and 3 months after treatment will be compared both within and between groups.

ELIGIBILITY:
Inclusion Criteria:

* Heel pain for at least 6 months consistent with clinical examination and imaging methods
* Numeric rating scale (NRS) in the first few steps in the morning ≥ 6
* Plantar fascia thicker than 4 mm as measured by ultrasonography
* Demonstration of calcaneal spur by X-ray
* Non-response to at least two of the indicated conservative treatments (rest, stretching exercises, oral anti-inflammatory drugs, silicone heel cup, local steroid injection, extracorporeal shock wave therapy (ESWT))

Exclusion Criteria:

* Achilles tendinopathy or calcaneal fracture
* Inflammatory or degenerative arthritis
* Spondyloarthropathies
* Tarsal tunnel syndrome (confirmed by electromyography if clinically suspected)
* Previous surgery on the plantar fascia or heel
* Diabetes mellitus, peripheral neuropathies, peripheral ischemic disease
* History of malignancy, pregnancy
* Anticoagulant-anticoaggregant drug use or coagulopathy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-08-05 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Numerical rating scale (NRS) | Change from baseline to 1st and 3rd month after treatment
  NRS is a scale that can be used measuring pain. Scores range from 0 (no pain) to 10 (the worst pain)

SECONDARY OUTCOMES:
The American Orthopedic Foot and Ankle Society (AOFAS) ankle hindfoot score | Change from baseline to 3rd month after treatment
  The AOFAS ankle-hindfoot score is used to measure the treatment outcome for ankle and hindfoot problems. It consists of three parts: pain, function, and alignment. Pain is worth 40 points, function is worth 50 points, and alignment is worth 10 points. The total score ranges from 0 to 100, with higher scores indicating better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Gevher Rabia Genc Perdecioğlu, Study Chair — Diskapi TRH
Locations (1):
- Diskapi Training and Research Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Yildiz G, Perdecioglu GRG, Yuruk D, Can E, Akkaya OT. Comparison of tibial nerve pulsed radiofrequency and intralesional radiofrequency thermocoagulation in the treatment of painful calcaneal spur and plantar fasciitis: a randomized clinical trial. Pain Med. 2024 Aug 1;25(8):493-499. doi: 10.1093/pm/pnae029. PMID 38652568